CLINICAL TRIAL: NCT03445091
Title: Open Label, Prospective Clinical Trial to Evaluate Impact on Quality of Life in Chronic Venous Insufficiency Patients Using SANKOM® Patent Socks During 4 Weeks
Brief Title: Study to Evaluate Impact SANKOM Patent Socks in Patients With CVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sankom SA (Industry)
Collaborators: InterMedService SA (Other); Pharmaxi LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Sankom-001
Record Dates: First submitted 2018-02-14; First posted 2018-02-26 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Chronic Venous Insufficiency
Keywords: compression socks; venous insufficiency; compression stockings; compression; compression therapy
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients using investigational product (Experimental): Open-label use of SANKOM Patent Socks
  Interventions: Device: SANKOM Patent Socks

INTERVENTIONS:
Device: SANKOM Patent Socks — Using compression socks to ease symptoms of patients with chronic venous insufficiency
  Other Names: gradient compression socks

SUMMARY:
Clinical study to evaluate impact on quality of life in patients with Chronic Venous Insufficiency during 4 weeks period of using SANKOM® Patent Socks

DETAILED DESCRIPTION:
Despite the application of compression stockings looks simple, it must be remembered that inappropriately worn stockings have the potential to cause certain problems. Unevenly distributed and excess pressure may break the skin, especially in older, malnourished patients and those with thin, brittle skin.

Although an extreme case, it highlights the importance of careful assessment, application, and monitoring of compression stockings.

Typically, the stockings are safe and wearing them results in few or no complications, provided they're worn smoothly against the leg, without any folds. But some groups of people should avoid them, including those with peripheral neuropathy or any other condition that impacts skin sensation; a history of a peripheral arterial bypass grafting; peripheral artery disease; skin infection; dermatitis with oozing or fragile skin; massive leg swelling; or pulmonary edema from congestive heart failure. Each of these conditions presents a different series of risks. For example, for people with peripheral artery disease, stockings can worsen oxygen delivery in arteries with impaired blood flow. People who have sensory problems, such as those with peripheral neuropathy, may not feel when a compression stocking is too tight, which could impede circulation. And certain skin conditions or infections may worsen with a compression stocking covering and pressing on the area.

In general, if subject has any medical condition, he/she should talk with health care professional before using compression stockings to see if they are good candidate for them.

Since probability of side/adverse effects from IP use is considered as very low vs of high probability of expected positive effects.

Study Purpose and Design Multi-center, observational open label study aimed to evaluate an impact on quality of life in Chronic Venous Insufficiency patients using SANKOM® Patent Socks during 4 weeks

This study will involve a maximum of 30 subjects. Subjects will be followed through outpatient's observation.

Primary Objective

Improvement of QoL by scores of:

* Aberdeen Varicose Veins Questionnaire (AVVQ)
* CIVIQ-2 Venous Quality of Life Questionnaire

Secondary Objectives

Secondary Endpoints are:

* Improvement of US-examination picture
* Improvement of QoL by Subject's questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Subject is informed and given ample time and opportunity to think about his/her participation and has given his/her written informed consent before any procedure;
2. Subject is male or female, 35-65 years of age;
3. Subject with chronic venous insufficiency CEAP (C1, C2);
4. Subject can speak and understand Ukrainian or Russian language.

Exclusion Criteria:

1. Subject participated in any clinical study (drug or device) within 6 months prior to the screening;
2. Subject unable to wear compression stockings;
3. Subject using other compression therapy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of health status in varicose veins patients | 4 weeks
  By mean of growing Aberdeen Varicose Veins Questionnaire score (total range 0 - 60). The higher values represent a better outcome.

SECONDARY OUTCOMES:
Improvement of Quality of Life | 4 weeks
  Growing of scrore of Quality of life questionnaire in Chronic Lower Limb Venous Insufficiency (CIVIQ-2) is expected
Improvement of ultara sound examination measures | 4 weeks
  Speed of venous blood flow of lower limbs is measured
Improvement of subject's self-assessment questionnaire | 4 weeks
  Subjective assessment of visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Serge M Mazourik, MD, Study Chair — Intermedservice
Locations (2):
- Ukraine (2):
  - Kyiv City Clinical Hospital No 6, Kyiv
  - Medical Consulting Center of Pechersk District, Kyiv

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the data yet.